CLINICAL TRIAL: NCT02445144
Title: Establishment of Functional MRI Imaging Parameters for Use in the Evaluation of Sickle Cell Disease
Status: Terminated | Type: Observational
Why Stopped: lack of funding
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Henny Billett, Chief, Division of Hematology, Department of Medicine, Albert Einstein College of Medicine
Other Study IDs: 2014-3574
Record Dates: First submitted 2015-04-15; First posted 2015-05-15 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Sickle Cell Anemia
Keywords: Inflammation; Blood Flow; Cognition
MeSH Terms: conditions — Anemia, Sickle Cell; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for evaluation of inflammatory markers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SCA Patients: Asymptomatic sickle cell anemia patients will undergo imaging/neurocognitive testing and be compared to controls
- Control Patients: Asymptomatic sickle cell anemia patients will undergo imaging/neurocognitive testing and be compared to controls

SUMMARY:
Patients with sickle cell anemia (SCA) are at an increased risk for damage to brain tissue due to their disease. The investigators are interested in how blood flow and cerebral inflammation are different in SCA patients and how that affects brain tissue- the investigators will use a relatively new set of dynamic MRI techniques to evaluate these parameters. The investigators will image participants with both SCA and matched controls with non-invasive MRI.

DETAILED DESCRIPTION:
Patients with sickle cell anemia (SCA) are at increased risk for episodes of stroke, both overt clinically evident and subclinical lesions only seen on imaging, which have associated morbidity and mortality. In addition, SCA patients demonstrate relatively poorer cognitive performance compared to their peers without SCA that is believed to be related to the episodes of stroke, but may be present even in their absence.

This study is designed to explore potential risk factors in patients with SCA that will identify predictors of cerebral damage that may also be modifiable. Elevated blood flow in cerebral arteries and increased inflammation are believed to be related to both ischemic lesions and cognitive findings but have not yet been clearly proven. We aim to use new MRI techniques which target cerebral blood flow and inflammation to identify differences in SCA patients and peers and follow this with an initial exploration of the association between these pathologic findings and cognitive deficits.

The investigator does not assign specific interventions to the subjects of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with HbSS/HbSB0,
* age between 18 and 55 years or age/gender/race/education matched peer

Exclusion Criteria:

* Previous history of a stroke/transient ischemic attack,
* neurosurgery,
* head trauma,
* seizures,
* pulmonary embolism,
* deep-vein thrombosis,
* bleeding/clotting disorders,
* current or previous use of anticoagulation medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 18-55 year old male and female patients with sickle cell anemia who are asymptomatic of previous CNS disease
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-11; Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow (CBF) measured by continuous arterial spin labeling (CASL) MRI | Day 1
  CBF will be measured by continuous arterial spin labeling (CASL) MRI

SECONDARY OUTCOMES:
Cogstate Testing | Day 1
  Exploration of the association between CBF values and cognitive performance deficits
Mean diffusivity/Fractional anisotropy (MD/FA) evaluated by diffusion tensor imaging (DTI) MRI measurements | Day 1
  MD/FA will be evaluated by diffusion tensor imaging (DTI) MRI measurements

CONTACTS AND LOCATIONS:
Overall Officials: Henny H Billett, MD, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center (Einstein), The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available after manuscript publication to those that request it
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Time frame of study has ended. Only preliminary data will be available - no end date
Access Criteria: Other investigators